CLINICAL TRIAL: NCT00203593
Title: EXercise for the Prevention of Syncope Evaluation
Brief Title: Exercise and Prevention of Syncope: EXPOSE
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: No Resources - No Personnel
Sponsor: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18413
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-03-14 (Estimated); Status verified 2007-03

CONDITIONS: Syncope
Keywords: exercise; total peripheral resistance; venoconstriction; blood volume expansion; orthostatic tolerance
MeSH Terms: conditions — Syncope; Motor Activity | interventions — Exercise; Blood Volume Determination; Lower Body Negative Pressure; Heart Rate; Blood Pressure; Vascular Resistance

INTERVENTIONS:
Behavioral: Exercise
Device: Blood volume
Procedure: VO2max test
Procedure: Lower body negative pressure
Behavioral: Heart Rate
Procedure: Blood Pressure
Behavioral: Total Peripheral Resistance

SUMMARY:
The purpose of this study is to determine whether eight weeks of exercise performed at an intensity of approximately 65% VO2max will improve symptoms associated with fainting (vasovagal syncope).

DETAILED DESCRIPTION:
Background: Vasovagal syncope affects 20-30% of the population, and for those who faint recurrently it causes a significant reduction in the quality of life. Although significant progress has been made in the past 15 years in our understanding of its diagnosis and prognosis, our therapeutic attempts often end in failure. Many patients who have been diagnosed with vasovagal syncope have a reduced orthostatic tolerance. Improved orthostatic tolerance has been achieved through exercise in a number of studies on healthy individuals. However, its efficacy as a means of treatment for those with vasovagal syncope has not been thoroughly explored.

Comparison: Subjects will be randomized to one of two groups: an exercise group or control. The exercise group will be asked to train at a target of approximately 65% of their maximum exercise capacity (VO2max) for 8 weeks/3 times per week. The control group will be asked to perform a series of neck rotation exercises. Orthostatic tolerance will be examined in both groups pre and post intervention.

ELIGIBILITY:
Inclusion Criteria: a diagnosis of vasovagal syncope as the cause of loss of consciousness, >1 lifetime syncope spell preceding enrolment, >-3 points on the S3 score for structurally normal hearts, >18 yrs of age with informed consent -

Exclusion Criteria: subjects with a negative Physical Activity Readiness Questionnaire (PARQ), those who are unable to provide informed consent, those with a VO2max >55ml/kg/min, those who exercise more than 30 minutes per day, 3 times per week, other causes of syncope, individuals with valvular, coronary, myocardial, or conductive abnormality, significant arrhythmia, hypertrophic cardiomyopathy, permanent pacemaker, seizure disorder, heart failure, major chronic cardiovascular disease, or renal dysfunction.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-03; Study Completion 2007-06

PRIMARY OUTCOMES:
Orthostatic tolerance - this will be measured at baseline and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Sheldon, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary (Health Sciences Center), Calgary, Alberta, Canada